CLINICAL TRIAL: NCT06553742
Title: High Definition Profiling of Ovarian Cancer Ascites for the Identification of Prognostic Biomarkers and Immunotherapeutic Targets: an Integrative Cell of Origin-guided Approach
Brief Title: High Definition Profiling of Ovarian Cancer Ascites
Status: Not yet recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: L2-016
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer; High Grade Ovarian Serous Adenocarcinoma; Ascites
MeSH Terms: conditions — Ovarian Neoplasms; Ascites

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 50 AS pre-chemotherapy samples will be collected at Istituto Europeo di Oncologia (IEO) AS samples will be centrifuged, lysis of red blood cells will be performed, and the cell pellet will be viable frozen. Frozen vials will be processed to isolate the tumor and non-immune tumor-associated cell populations (CD45-), or gradient separation to isolate immune cells.
  The CD45- population will be used for:
  i) genomic DNA extraction that will be subjected to DNA methylation profiling (EPIC 850k arrays, Illumina) and origin-based stratification.
  ii) generation of sMOCS, that allow to enrich for cancer stem cells, through label-free FACS sorting into 96-well low attachment plates.
  iii) single cell transcript profiling of both CD45- cells and dissociated sMOCS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project entails the collection of a prospective cohort of ascites (AS) samples from High Grade Serous Ovarian Cancer (HGSOC) patients.

High Grade Serous Ovarian Cancer (HGSOC) is a major cause of cancer-related mortality, due to the late-stage diagnosis and failure of surgery and chemotherapy (CHT) to eradicate the disease with no significant improvement in overall survival.

The primary objective of the project is to generate a comprehensive map of ascites cell components, detailing both their intrinsic features and the landscape of cellular interactions mediated by soluble factors in ascitic fluid.

DETAILED DESCRIPTION:
HGSOC is a major cause of cancer-related mortality, due to the late-stage diagnosis and failure of surgery and chemotherapy (CHT) to eradicate the disease with no significant improvement in overall survival.

In recent years, new therapeutic regimens are being tested to improve the care of HGSOC patients. These approaches include the use of poly-ADP-ribose polymerase inhibitors (PARPi) targeting Homology Directed Repair deficiency, anti-angiogenic drugs, such as anti-VEGF monoclonal antibodies, and immune checkpoint inhibitors, that target immune modulation induced by tumor and tumor-associated cells and inflammatory signals. Unfortunately, the outcome of such therapies has been to date either erratic or dismal.

This points to the acute need to identify new biomarkers predictive of treatment response, effectively geared to the clinical setting.

The primary objective of the project is to generate a comprehensive map of ascites cell components, detailing both their intrinsic features and the landscape of cellular interactions mediated by soluble factors in ascitic fluid. This will allow to define tumoral archetypes, reflecting HGSOC's endophenotypes, associated with prognosis in patients, possibly guiding future refined therapeutical paradigms for ovarian cancer patients and endowing researchers with a well-characterized multilayered dataset for future reference in the context of molecular dissection and target discovery paradigms.

Indeed, the combination of origin- and archetype-based stratification of HGSOC patients, will allow to better identify patients for which existing therapeutical regimens could be beneficial, such as the use of checkpoint inhibitors and anti-angiogenic drugs, that have been so far erratic in ameliorating patient's survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicious or confirmed ovarian cancer pathology undergoing debulking surgery
* Diagnosis of high grade serous ovarian cancer confirmed by histopathology assessment
* Patients who provided written informed consent

Exclusion Criteria:

* HIV-positive patients
* HBV-positive patients
* HCV-positive patients

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: HGSOC samples are provided by the European Institute of Oncology biobank. All patients will be provided written informed consent.
  Patients with suspicious or confirmed ovarian cancer pathology undergoing debulking surgery will be included in the protocol. Only samples diagnosed as high grade serous ovarian cancer confirmed by histopathology assessment will be included in the following analyses.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Generation of a comprehensive map of ascites cell components | 48 month
  The samples will be stratified according to a DNA-methylation based signature specific for the tissue of origin of HGSOC.
  The cellular fraction derived from ascites samples will be profiled by single cell multiomics to define the cell populations associated to either the fallopian tube or ovarian surface epithelium origin. In parallel, ascitic fluid will be profiled by ELISA to define the soluble components present in the two HGSOC subtypes. These data will be used to generate a map of ascites cell components and biomarkers specific for the two tissues of origin of this disease. This map will be exploited to highlight possible therapeutic avenues for HGSOC patients.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Testa, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy